CLINICAL TRIAL: NCT04421183
Title: Investigation of the Serum MUC3 Protein Levels in Gestational Hypertensive Disease (Preeclampsia-Eclampsia, Pregnancy Induced Hypertension, and HELLP Syndrome) Compared With Normal Pregnancy
Brief Title: Investigation of the Serum Mucoprotein 3 (MUC3) Protein Levels in Gestational Hypertensive Disease
Acronym: MUC3
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Guven, professor, Karadeniz Technical University
Other Study IDs: MUC 3
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Muc3; Pregnancy Induced Hypertension
Keywords: Muc3; Preeclampsia; Eclampsia; HELLP
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: preeclampsia
  Interventions: Diagnostic Test: draw blood
- 4: normal pregnancy without complication
  Interventions: Diagnostic Test: draw blood
- 2: hellp
  Interventions: Diagnostic Test: draw blood
- 3: eclampsia
  Interventions: Diagnostic Test: draw blood

INTERVENTIONS:
Diagnostic Test: draw blood — draw blood from the all of patients

SUMMARY:
Hypertensive diseases of pregnancy are one of the most frequently encountered reasons for maternal and neonatal morbidity and mortality. The excretion of high levels of mucoprotein takes part in the pathogenesis of preeclampsia through restraining trophoblast invasion. This study aimed to investigate levels of serum mucoprotein three in hypertensive diseases of pregnancy. This study included a total of eighty cases that 20 normal pregnancy, 20 gestational hypertension, 20 preeclampsia, and 20 HELLP syndrome patients from June 2010- January 2011.

DETAILED DESCRIPTION:
Hypertensive diseases of pregnancy are one of the most frequently encountered reasons for maternal and neonatal morbidity and mortality. The excretion of high levels of mucoprotein takes part in the pathogenesis of preeclampsia through restraining trophoblast invasion. This study aimed to investigate levels of serum mucoprotein three in hypertensive diseases of pregnancy. This study included a total of eighty cases that 20 normal pregnancy, 20 gestational hypertension, 20 preeclampsia, and 20 HELLP syndrome patients from June 2010- January 2011. This is the first study measuring levels of serum mucoprotein three in gestational hypertensive disease. MUC3 levels showed a distinctive increase in hypertensive diseases of pregnancy compared with the pregnant control group. As a result, it is found that plasma mucoprotein 3 levels increase as the severity of hypertensive diseases of pregnancy increases; and plasma mucoprotein 3 could be a precursor for the evaluation of the severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

* To accept the consent to participate in the research and sign the form,
* According to ACOG 2002, pregnancy meets the criteria of hypertensive diseases [1], The diagnosis of HELLP syndrome was made according to the criteria described by Sibai. These; abnormal peripheral smear, schistocyte in the peripheral smear, lactate dehydrogenase > 600 U / L, hemolysis, total bilirubin> 1.2 mg / dl, AST> 70 U / L, platelet count <100,000mm3.
* When the demographic characteristics and CVs of all cases were questioned in the initial evaluation, not having chronic inflammation or acute infection, not having any systemic disease, recurrent pregnancy loss, thrombophilia, antiphospholipid antibody syndrome,
* Not smoking, No history of cancer, No multiple pregnancies
* Not using antihypertensive, anticoagulant, NSAID, corticosteroid or antiplatelet and antiepileptic drugs

Exclusion Criteria:

* using antihypertensive, anticoagulant, NSAID, corticosteroid or antiplatelet and antiepileptic drugs
* smoking,history of cancer, multiple pregnancies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy is female-specific. therefore, women were included in the study.
Study Population: patients who were diagnosed with hypertensive disease among the patients who applied to the pregnant clinic of Karadeniz Technical University Faculty of Medicine, Obstetrics and Gynecology Department with the approval of the KTÜ Faculty of Medicine Research Ethics Committee dated 27.05.2010 and 154 number ( 80 cases, including the study group and 20 normotensive pregnant control group) were included in the study between June 2010 and January 2011.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2011-01-01 (Actual); Study Completion 2011-01-02 (Actual)

PRIMARY OUTCOMES:
Collection of Blood Samples | 6 months
  The blood samples required for the study were obtained from samples taken into a heparinized tube. Maternal blood samples were taken at the time of diagnosis in patients with preeclamptic - eclamptic, gestational hypertension and HELLP syndrome before starting any treatment when they apply for delivery in normal pregnant women. After the blood samples were centrifuged at Eppendorf Centrifuge-5084R at 3000 G for 10 minutes, the serum was separated. Some of the serum collected were placed in a 1.5 cc Eppendorf tube and stored at -80 ˚C in the medical cooler (Ariston) in the Department of Obstetrics and Gynecology.
Measurement of Mucoprotein in Serum | 1 month
  After collecting all serum samples (80 pieces), they were dissolved at room temperature and MUC3 (Human Mucin 3, MUC3 ELISA Kit) level was measured in serum samples with the help of commercial ELISA kits. The measurement technique principle is given below.Mucoprotein content in serum was determined in ng/ml with the help of a special ELISA kit system and elements for mucoprotein 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technique University, Trabzon, Ortahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No